CLINICAL TRIAL: NCT06973538
Title: Is Music-Enhanced Calisthenic Exercise More Effective in Healthy Sedentary Older Adults?
Brief Title: Music-Enhanced Calisthenics in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Feyza Altindal Karabulut (Other)
Responsible Party: Sponsor-Investigator, Feyza Altindal Karabulut, Assistant Professor, Nigde Omer Halisdemir University
Organization: Nigde Omer Halisdemir University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/7-5
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Balanced; Quality of Life; Exercise Theraphy; Proprioception

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model in which participants are randomly assigned to one of three independent groups:
  Music-based Calisthenic Exercise Group (MCEG): Participants perform calisthenic exercises with background music.
  Calisthenic Exercise Group (CEG): Participants perform the same exercises without music.
  Control Group (CG): Participants receive no structured exercise intervention.
  Each group follows a fixed 8-week intervention program, with sessions conducted twice weekly. The primary aim is to assess the effects of music-enhanced calisthenic exercises on balance, muscle strength, proprioception, and quality of life in healthy sedentary older adults. Data will be collected pre- and post-intervention to evaluate the effectiveness of the interventions. Randomization ensures that each participant has an equal chance of being assigned to any of the three groups, reducing selection bias and enhancing the internal validity of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Music-based Calisthenic Exercise Group (MCEG) (Experimental): Participants in this group will perform calisthenic exercises with background music for 8 weeks. Each session will include a 10-minute warm-up, 30 minutes of music-enhanced calisthenic exercises (e.g., seated leg lifts, chair squats, seated marching, arm curls, and seated torso twists), and a 10-minute cool-down. From the fifth week onwards, elastic resistance bands will be introduced to progressively increase exercise intensity. The music selection is designed to promote engagement and motivation, including rhythmic and motivational tracks suitable for older adults.
  Interventions: Other: Music-based Calisthenic Exercise
- Arm 2: Calisthenic Exercise Group (CEG) (Experimental): Participants in this group will perform the same calisthenic exercises as the MCEG but without background music. The intervention will last 8 weeks, with each session including a 10-minute warm-up, 30 minutes of calisthenic exercises (e.g., seated leg lifts, chair squats, seated marching, arm curls, and seated torso twists), and a 10-minute cool-down. From the fifth week onwards, elastic resistance bands will be introduced to progressively increase exercise intensity.
  Interventions: Other: Music-based Calisthenic Exercise
- Arm 3: Control Group (CG) (No Intervention): Participants in this group will not receive any structured exercise intervention during the 8-week study period. They will be encouraged to maintain their usual daily activities without any specific exercise regimen. This group serves as a baseline for comparison against the exercise groups.

INTERVENTIONS:
Other: Music-based Calisthenic Exercise — Participants in this group will perform 8 weeks of calisthenic exercises with background music. Each session includes a 10-minute warm-up, 30 minutes of music-based exercises (e.g., seated leg lifts, chair squats, arm curls), and a 10-minute cool-down. Elastic resistance bands will be introduced from week 5 to increase intensity. Music tracks are selected to enhance motivation and engagement.
  Other Names: Calisthenic Exercise
  Arms: Arm 1: Music-based Calisthenic Exercise Group (MCEG); Arm 2: Calisthenic Exercise Group (CEG)

SUMMARY:
This study aimed to evaluate the effects of music-enhanced calisthenic exercises on balance, muscle strength, proprioception, and quality of life (QoL) in sedentary older adults. Thirty-one participants (mean age: 74.41 ± 5.86 years) were randomly assigned to three groups: Calisthenic Exercise Group (CEG), Music-based Calisthenic Exercise Group (MCEG), and Control Group (CG). The intervention consisted of 16 sessions over 8 weeks, including a 10-minute warm-up, 30 minutes of exercise, and a 10-minute cool-down. Assessments included the Timed Up and Go Test (balance), Sit-to-Stand Test (strength), joint position sense tests (proprioception), and the Nottingham Health Profile (QoL). Both exercise groups showed significant improvements in all measured outcomes (p<0.05), with the MCEG demonstrating superior gains, particularly in energy levels and physical function. These findings support the use of music to enhance the benefits of exercise in older adults.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) aimed to evaluate the effects of music-enhanced calisthenic exercises on balance, muscle strength, proprioception, and quality of life (QoL) in healthy sedentary older adults living in nursing homes. The study included 31 participants aged 65 years and older, randomly assigned to one of three groups: the Calisthenic Exercise Group (CEG), the Music-based Calisthenic Exercise Group (MCEG), and the Control Group (CG). The intervention was conducted over 8 weeks, consisting of 16 sessions, with each session lasting approximately 50 minutes. Sessions included a 10-minute warm-up, 30 minutes of calisthenic exercises, and a 10-minute cool-down. The MCEG performed the exercises with background music, while the CEG performed the same exercises without music. The CG did not receive any structured exercise intervention.

The calisthenic exercises included seated leg lifts, chair squats, seated marching, arm curls, and seated torso twists. From the fifth week onwards, elastic resistance bands were introduced to progressively increase the difficulty level and promote muscle hypertrophy and strength gains. Music tracks for the MCEG were carefully selected to promote engagement and motivation, including popular rhythmic and motivational songs suitable for older adults.

Assessments were conducted pre- and post-intervention using standardized measurement tools. Balance was assessed using the Timed Up and Go (TUG) Test, muscle strength with the Sit-to-Stand Test, proprioception with joint position sense testing, and quality of life with the Nottingham Health Profile (NHP). These assessments were chosen to capture the physical and psychological impact of the exercise interventions, providing a comprehensive evaluation of the participants' physical function and overall well-being.

Data were analyzed using SPSS (v22.0), with parametric or non-parametric tests selected based on data distribution. Paired t-tests or Wilcoxon signed-rank tests were used for within-group comparisons, while ANOVA or Kruskal-Wallis tests were applied for between-group comparisons. A p-value of <0.05 was considered statistically significant.

Ethical approval for the study was obtained from the Non-Interventional Ethics Committee of Niğde Ömer Halisdemir University (Approval No: 2022/11-12, dated 26.09.2022). All participants provided written informed consent before participating in the study.

The primary aim of this study was to determine whether music-enhanced calisthenic exercises provide greater physical and psychological benefits compared to standard calisthenic exercises alone. Secondary aims included evaluating changes in balance, muscle strength, proprioception, and overall quality of life among healthy sedentary older adults. The results are expected to provide evidence supporting the use of music as a simple, low-cost, and enjoyable addition to exercise programs for older adults.

ELIGIBILITY:
Inclusion Criteria:

Only individuals deemed physically suitable for exercise by the institutional physician and who agreed to participate in the exercise program were included.

Exclusion Criteria:

Individuals under 65 years of age.

Severe cognitive impairment or diagnosed dementia that would prevent safe participation in the exercise program.

Severe musculoskeletal, neurological, or cardiovascular conditions that contraindicate physical exercise.

Acute or unstable medical conditions requiring immediate medical intervention.

Hearing impairment that would significantly reduce the ability to follow music-based exercises.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Balance Improvement | Baseline and 8 weeks post-intervention
  Change in balance as measured by the Timed Up and Go (TUG) Test. This test assesses functional mobility and balance, with a shorter completion time indicating better balance. Lower TUG scores at the end of the 8-week intervention indicate improved balance.
  Change in balance as measured by the Timed Up and Go (TUG) Test. This test assesses functional mobility and balance, with a shorter completion time indicating better balance. Lower TUG scores at the end of the 8-week intervention indicate improved balance.
Muscle Strength Improvement | Baseline and 8 weeks post-intervention
  Change in lower limb muscle strength as measured by the Sit-to-Stand Test. This test counts the number of full stands a participant can perform in 30 seconds. Higher scores indicate better muscle strength.
Proprioception Improvement | Baseline and 8 weeks post-intervention
  Change in joint position sense as measured by the Joint Position Sense Test. Smaller deviations from the target angle indicate better proprioceptive function.
Quality of Life (QoL) Improvement Quality of Life (QoL) Improvement | Baseline and 8 weeks post-intervention
  Change in quality of life as measured by the Nottingham Health Profile (NHP), which assesses physical mobility, emotional reactions, social isolation, pain, and energy levels. Lower NHP scores indicate better perceived quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Ömer Halisdemir University, Faculty of Health Sciences, Niğde, Ni̇ğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data, including demographic information, Timed Up and Go (TUG) test scores, Sit-to-Stand test results, joint position sense measurements, and Nottingham Health Profile (NHP) scores, will be made available upon reasonable request. Data will be shared through a secure institutional repository following publication of the primary manuscript. Access will be granted to qualified researchers for the purpose of validating findings or conducting further analysis, in accordance with ethical guidelines.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Baseline (Pre-intervention) and 8 weeks post-intervention